CLINICAL TRIAL: NCT02189512
Title: CD14/CD16 Activation in Brain-death Organ Donors and Effect of Surgical Intestinal Manipulation
Brief Title: Study on the Effect of Surgical Intestinal Manipulation
Acronym: IMMO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IMMO-20140206
Record Dates: First submitted 2014-05-27; First posted 2014-07-14 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-05

CONDITIONS: Intestinal Manipulation
Keywords: brain-death organ donors; intestinal manipulation; monocytes
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- brain death organ donors (Other): cases - blood sampling
  Interventions: Other: blood sampling
- abdominal aortic aneurysm repair (Other): controls - blood sampling
  Interventions: Other: blood sampling

INTERVENTIONS:
Other: blood sampling — cases - blood sampling controles - blood sampling

SUMMARY:
The aim of this study is to study the impact of brain death and surgical small bowel manipulation on the release of different types of monocytes.

ELIGIBILITY:
Inclusion Criteria:

* patients who are brain death
* patients who undergo an elective abdominal aortic aneurysm repair

Exclusion Criteria:

* < 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-05; Primary Completion 2016-01 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
subtypes of monocytes | 1 day
  evaluate different subtypes of monocytes in brain-death donors by collecting portal and peripheral blood after lapaotomy and before dissection
evaluate effect of intestinal manipulation | 1 day
  evaluate the effect of intestinal manipulation on the different subtypes of monocytes and pro-/anti-inflammatory cytokines

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Pirenne, MD,PhD, Principal Investigator — Abdominal Transplant Surgery, University Hospitals Leuven, KULeuven
Locations (1):
- University Hospitals Leuven, Leuven, Vlaams-Brabant, Belgium